CLINICAL TRIAL: NCT04575493
Title: Clinical Efficacy of Crano-cure inTreatment of Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamia University of Bahawalpur (Other)
Collaborators: Hamdard University (Other)
Responsible Party: Principal Investigator, Hafiz Abdul Sattar Hashmi, Principal Investigator, Islamia University of Bahawalpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EM-DP-14-001
Record Dates: First submitted 2020-09-25; First posted 2020-10-05 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Clinical trials are designed to understand the nature of disease, its associated symptoms, and patient's response towards management. The study has aim to evaluate the effect of medical intervention with allopathic and herbal medicine to treat urinary tract infection. For this purpose, the patient suffering from urinary tract infection were examined and managed in different medical centers such as Shifa-ul-Mulk Memorial Hospital Hamdard University Karachi, Naseem ul Sehat Eastern Medicine Clinic Bahawalpur, Matab Hakeem Atta ur Rehman Siddique Lahore and khurshid Siddique Clinic Lahore.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): No of enrolled Pts. 102 Drug Cap. Crano-cure 500mg. Quantity 500 mg Bd Usage 1 cap Bd Duration of study 14 days Follow up 1st follow up after 2 weeks 2nd follow up after 4 weeks
  Interventions: Dietary Supplement: Crano-cure
- control group (Active Comparator): No of enrolled Pts. 103 Drug Tab. Ciprofloxacin 500mg Quantity 500mg Bd Usage 1 Tab Bd Duration of study 14 days Follow up 1st follow up after 2 weeks 2nd follow up after 4 weeks
  Interventions: Drug: Ciprofloxacin 500 mg

INTERVENTIONS:
Dietary Supplement: Crano-cure — Research literatures have revealed that Tribulus terrestris (Gokhro), Vaccinium macrocarpon (karonda), Cuminum cyminum (Zeera sufaid), Rheum emodi (Revand chini) and Piper cubeba (Kabab chini) are important therapeutic plants. Many pharmacological researches have been done on these plants. For instance, antioxidant, antiseptic, anti-microbial, anti-bacterial, anticancer etc. In the above claims and facts, the study is conducted to formulate and evaluate the polyherbal capsule and to find out the most effective combination having anti-bacterial activity.
  Arms: Test Group
Drug: Ciprofloxacin 500 mg — Being a standard drug as antibiotic and will be used in Control group.
  Arms: control group

SUMMARY:
The main objectives of the study are; to determine the efficacy of test drug Crano-cure for the treatment of urinary tract infection, to compare the effectiveness of Polyherbal formulation Crano-cure vs. Standard allopathic. Antibacterial/ antibiotic (Ciprofloxacin 500 mg) in treatment of UTI, to assess the safety of trial drug.

Research literatures have revealed that Tribulus terrestris (Gokhro), Vaccinium macrocarpon (karonda), Cuminum cyminum (Zeera sufaid), Rheum emodi (Revand chini) and Piper cubeba (Kabab chini) are important therapeutic plants. Many pharmacological researches have been done on these plants. For instance, antioxidant, antiseptic, anti-microbial, anti-bacterial, anticancer etc. In the above claims and facts, the study is conducted to formulate and evaluate the polyherbal capsule and to find out the most effective combination having anti-bacterial activity.

DETAILED DESCRIPTION:
A urinary tract infection (UTI) is the infection of kidney that affects urinary tract. It affects the urinary bladder (cystitis) and kidney (pyelonephritis). Symptoms of urinary bladder infection are painful urination, frequent micturation, and urinary incontinence. Symptoms of infection in kidney include pyrexia and lumber pain also in addition to symptoms of a lower urinary tract infection and rarely blood in the urine. In older age and in young adults, symptoms may be unclear or non-specific [1].

Urinary tract infections are grouped into two types; complicated and uncomplicated. In uncomplicated cases of urinary tract infections, the function of urinary tract system does not disturb. In complicated UTI, the normal function of UT system disturbs [2].

Uncomplicated UTI is usually caused by E. coli Staphylococcus saprophyticus Klebsiella pneumonia Proteus mirabilis Enterococcus spp. While complicated UTI is caused by Similar organisms which causes uncomplicated UTI Staphylococcus spp. Enterococcus spp. P. aeruginosa

Current studies on the prevalence of urinary tract infections approximately one third population of the world has been suffering from this disease. This disease causes Pyuria, burning urination, heamaturia, pyrexia, Vaginal itching, Offensive" smell and turbid urine, urinate frequent, urgency to urinate and suprapubic pain or pain in pelvis. It is not life-threatening disease. Different antibacterial/ antibiotics are available such as Co-trimaxazole, amoxicillin, nitrofurantoin, trimethoprim, combination of trimethoprim and sulfamethoxazole and quinolone antibiotics is taken as a choice for the treatment of UTI [3]. The antibacterial agents/ antibiotic available but they are limited in number, have adverse effects, resistance of bacteria to these agents and relapse of the UTI. In order to overcome the problem of less availability of drugs needed to treat urinary tract infection, with traditional medicine derived from medicinal plants. This encouraged the search for new and dynamic antibacterial agents from plant sources.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 60 years with symptomatic acute urinary tract infection.

  * Willing to participate in the study
  * Non-pregnant adult females.
  * Clinical signs and symptoms of a UTI (e.g., dysuria, frequency, urgency to urinate, Burning sensations during urination, Hematuria, suprapubic pain) with onset of symptoms < 72 hours prior to study entry.
  * One positive pre-treatment clean-catch midstream urine culture within 48 hours of enrollment in the study, defined as > 105 CFU/mL.
  * Patients having all socioeconomic classes including lower, middle and higher.
  * In-vitro susceptibility testing of the uropathogen to test and control drug.

Exclusion Criteria:

* • Women who are pregnant, nursing, or not using a medically accepted, effective method of birth control. If an antimicrobial agent is to be studied for the treatment of UTI in pregnant women, this proposal should be justified, the risk/benefit expectations explained, and the issue presented to the division.

  * Three or more episodes of acute uncomplicated UTI in the past 12 months.
  * Patients with evidence of factors predisposing to the development of urinary tract infections, including calculi, stricture, primary renal disease (e.g., polycystic renal disease), or neurogenic bladder.
  * Patients with onset of symptoms 96 hours or more prior to entry.
  * Patients with a temperature > 1010 F, flank pain, chills, or any other manifestations suggestive of upper urinary tract infection.
  * Patients with known or suspected hypersensitivity to the test or control drug.
  * Patients who received treatment with other antimicrobials within 48 hours prior to entry.
  * Patient suffering in chronic illness Diabetes mellitus, chronic liver diseases

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 205 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Urine Culture Examination | 15 days
  Urine Culture examination for
  Escherichia coli Staphylococcus saprophyticus Klebsiella pneumonia Proteus mirabilis

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Jalil Ur Rehman, Bahawalpur, Punajb
  - University College of Conventional Medicine, Bahawalpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ur Rehman J, Iqbal A, Asif HM, Hadi F, Ahmed K, Ahmed M, Sumreen L. Alternative Approaches for the Management of Urinary Tract Infection with Crano-cure: A Randomized Clinical Trial. Altern Ther Health Med. 2024 Jul;30(7):12-19. PMID 39110045